CLINICAL TRIAL: NCT05307016
Title: Dilemma of the Appropriate Surgical Intervention of Morbidly Adherent Placenta: Could it be Solved Prenatally?
Brief Title: Morbidly Adherent Placenta, Diagnosis and Proper Management
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hatem Awaga, Lecturer of Obstetrics and Gynecology, Sohag University
Other Study IDs: Soh-Med-22-01-35
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Morbidly Adherent Placenta
Keywords: ultrasonography; Intraoperative staging; Histopathological assessment
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MAP patients: All pregnancies complicated with any degree of Placenta previa anterior, posterior or centralis undergoing pre-labor CS at gestational age (36+0 to 40+0)
  Interventions: Diagnostic Test: Two dimensional ultrasonography power and color doppler

INTERVENTIONS:
Diagnostic Test: Two dimensional ultrasonography power and color doppler — transabdominal and transvaginal two-dimensional power Doppler ultrasound volumes of the placental bed were obtained according to a predefined protocol with the participant in a semi-recumbent position and a full bladder using a RAB4-8-D 3D/4D curved array abdominal transducer (4-8.5 MHz) on a Voluson E8. Predetermined machine settings were used. To allow for differences in attenuation of the power Doppler signal resulting from variation in placental site and maternal adiposity.
  Intraoperative staging of degree of placental invasion will be done according to clinical grading system by Collins et al., 2015.
  Specimens obtained from patients who underwent hysterectomy or resection of segment of anterior uterine wall in cases with anterior placenta previa will be immersed in formalin 10% concentration and will be sent for histopathological evaluation that will be done by the same pathologist.
  Other Names: Intra-operative clinical staging during routine cesarean section of cases; postoperative histopathological assessment of available specimens

SUMMARY:
The main idea of this study is to establish the diagnostic criteria for cases of morbidly adherent placenta (MAP) using different ultrasonographic modalities and compare this with intra-operative findings and postoperative histopathological assessment

DETAILED DESCRIPTION:
This study is a clinical trial that will include all patients fulfilling the eligibility criteria and presented to the emergency unit of the department of Obstetrics and Gynecology in Sohag University hospital (Egyptian tertiary referral hospital) between February 2022 and February 2023. The attending physician will explain the nature of the study and all patients will be asked to sign an informed consent. A senior physician will evaluate the patient to confirm the diagnosis of placenta previa and degree of invasion in query accreta patients by using transabdominal and transvaginal US (Voluson,p8). 2D gray scale ultrasound, color and power doppler ultrasound will be performed firstly followed by 3D ultrasound.

All data will be saved in closed excel sheet and patients will be operated by a different surgical team, intraoperative staging of degree of placental invasion will be done according to clinical grading system by Collins et al., 2015 [5] in addition to histopathological evaluation when available, such as in cases of hysterectomy and cases with anterior placenta who were treated by excision of part of anterior uterine wall suitable for histopathological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* o All pregnancies complicated with any degree of Placenta previa anterior, posterior or centralis undergoing pre-labor CS at gestational age (36+0 to 40+0), patients will be divided into subgroups according to number of previous CS, presence or absence of antepartum hemorrhage and qualifications of operative theatre in previous deliveries (public or private sector).

Exclusion Criteria:

* Women with history of medical co-morbidities such as chronic hypertension, Diabetes mellitus, renal diseases, autoimmune diseases, history of organ transplantation and immunosuppressive therapy, hematological diseases, history of thrombotic events, cardiopulmonary diseases, liver diseases Acute and chronic inflammatory diseases.
* Pregnancy induced medical disorders like: Gestational hypertension, preeclampsia, Gestational diabetes, Gestational thrombocytopenia and proteinuria.
* Fetal anomalies.
* Emergency CS if the patient is in labor.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presented to the department of Obstetrics and Gynecology in Sohag University hospital between February 2022 and February 2023 complicated with any degree of Placenta previa undergoing pre-labor CS at gestational age (36+0 to 40+0),. The attending physician will explain the nature of the study and all patients will be asked to sign an informed consent. A senior physician will evaluate the patient to confirm the diagnosis of placenta previa and degree of invasion in query accreta patients by using transabdominal and transvaginal US (Voluson,p8).
  All data will be saved in closed excel sheet and patients will be operated by a different surgical team, intraoperative staging of degree of placental invasion will be done according to clinical grading system by Collins et al., 2015 in addition to histopathological evaluation when available.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Acurray of ultrasonographic features for diagnosis of different degrees of MAP | All pregnancies complicated by any degree of placenta previa undergoing pre-labor CS at gestational age (36+0 to 40+0) weeks
  The sensitivity and specificity of the ultrasonographic findings of MAP according to the final intraoperative diagnosis and available histopathological data

SECONDARY OUTCOMES:
The validity of ultrasonographic findings of MAP for selecting the appropriate surgical intervention | All pregnancies complicated by any degree of placenta previa undergoing pre-labor CS at gestational age (36+0 to 40+0) weeks
Evaluating the accuracy of this criteria in all types of placenta previa | All pregnancies complicated by any degree of placenta previa undergoing pre-labor CS at gestational age (36+0 to 40+0) weeks
Studying all factors that may affect the accuracy of this criteria such as number of previous CS, qualifications of the previous CS, presence or absence of antepartum hemorrhage. | All pregnancies complicated by any degree of placenta previa undergoing pre-labor CS at gestational age (36+0 to 40+0) weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Medical school, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gielchinsky Y, Rojansky N, Fasouliotis SJ, Ezra Y. Placenta accreta--summary of 10 years: a survey of 310 cases. Placenta. 2002 Feb-Mar;23(2-3):210-4. doi: 10.1053/plac.2001.0764. PMID 11945088
- [Background] Publications Committee, Society for Maternal-Fetal Medicine; Belfort MA. Placenta accreta. Am J Obstet Gynecol. 2010 Nov;203(5):430-9. doi: 10.1016/j.ajog.2010.09.013. PMID 21055510
- [Background] Jauniaux E, Collins SL, Jurkovic D, Burton GJ. Accreta placentation: a systematic review of prenatal ultrasound imaging and grading of villous invasiveness. Am J Obstet Gynecol. 2016 Dec;215(6):712-721. doi: 10.1016/j.ajog.2016.07.044. Epub 2016 Jul 26. PMID 27473003
- [Background] Palacios Jaraquemada JM, Bruno CH. Magnetic resonance imaging in 300 cases of placenta accreta: surgical correlation of new findings. Acta Obstet Gynecol Scand. 2005 Aug;84(8):716-24. doi: 10.1111/j.0001-6349.2005.00832.x. PMID 16026395
- [Background] Collins SL, Stevenson GN, Al-Khan A, Illsley NP, Impey L, Pappas L, Zamudio S. Three-Dimensional Power Doppler Ultrasonography for Diagnosing Abnormally Invasive Placenta and Quantifying the Risk. Obstet Gynecol. 2015 Sep;126(3):645-653. doi: 10.1097/AOG.0000000000000962. PMID 26214694
- [Background] Collins SL, Stevenson GN, Noble JA, Impey L, Welsh AW. Influence of power Doppler gain setting on Virtual Organ Computer-aided AnaLysis indices in vivo: can use of the individual sub-noise gain level optimize information? Ultrasound Obstet Gynecol. 2012 Jul;40(1):75-80. doi: 10.1002/uog.10122. PMID 22009687
- [Background] Hecht JL, Baergen R, Ernst LM, Katzman PJ, Jacques SM, Jauniaux E, Khong TY, Metlay LA, Poder L, Qureshi F, Rabban JT 3rd, Roberts DJ, Shainker S, Heller DS. Classification and reporting guidelines for the pathology diagnosis of placenta accreta spectrum (PAS) disorders: recommendations from an expert panel. Mod Pathol. 2020 Dec;33(12):2382-2396. doi: 10.1038/s41379-020-0569-1. Epub 2020 May 15. PMID 32415266